CLINICAL TRIAL: NCT00916253
Title: Method of Assessment of Driving Ability in Patients Suffering From Wakefulness Pathologies, Impact of Modafinil Treatment.
Brief Title: Method of Assessment of Driving Ability in Patients Suffering From Wakefulness Pathologies
Acronym: AUTOSOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: CHUBX 2008/37
Record Dates: First submitted 2009-05-29; First posted 2009-06-09 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Narcolepsy; Hypersomnia
Keywords: Sleep; real driving; simulated driving; MWT
MeSH Terms: conditions — Narcolepsy; Disorders of Excessive Somnolence | interventions — Modafinil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Modafinil First (Experimental): Treatment by Modafinil during first condition then placebo during second condition
  Interventions: Drug: Modafinil; Drug: Placebo
- Placebo First (Experimental): Treatment by Placebo during first condition then Modafinil during second condition
  Interventions: Drug: Modafinil; Drug: Placebo
- H (No Intervention): Healthy Volunteers

INTERVENTIONS:
Drug: Modafinil — Modafinil is taken by narcoleptics or hypersomniacs during 5 successive days, twice a day (at the breakfast and at the lunch):
  * during 3 days at home
  * during the period of 2 nights and 2 successive days of hospitalization in order to realise a Maintenance of Wakefulness Test the first day and 2 driving sessions (one simulated driving during the morning and one real driving during the afternoon) of 2 hours each the day after, under treatment (Modafinil).
  Arms: Modafinil First; Placebo First
Drug: Placebo — Placebo is taken by narcoleptics or hypersomniacs during 5 successive days, twice a day (at the breakfast and at the lunch):
  * during 3 days at home
  * during the period of 2 nights and 2 successive days of hospitalization in order to realise a Maintenance of Wakefulness Test the first day, and 2 driving sessions ( one simulated driving during the morning and one real driving during the afternoon) of 2 hours each the day after, under Placebo.
  Arms: Modafinil First; Placebo First

SUMMARY:
The project will improve scientific knowledge regarding a recent law applying potentially to every french driver. It will give for the first time an indication on the impact of alerting treatments on driving risks. It will reinforce the links between different research environments (sleep physiopathology, clinical research, cognitive neurosciences, driver's supervision, virtual reality, pharmacology) among the RESAT network (Réseau Eveil Sommeil Attention Transport). It will stimulate data acquisition in technological research to better understand the difference between real and simulated driving

DETAILED DESCRIPTION:
Excessive daytime sleepiness is responsible of 20% of traffic accidents and 2/3 of truck accidents on French Freeways. Since the publication of a new law (arrêté du 28 décembre 2005 du journal officiel) regulating fitness to drive, the Maintenance of Wakefulness Test (MWT) is now mandatory to evaluate driving skills of patients suffering of excessive daytime sleepiness. The MWT has shown a good predictability of driving handicap on simulators in patients suffering from obstructive sleep apnea syndrome. Nevertheless no study has proven yet the predictability of the MWT regarding real and simulated driving in narcoleptics and hypersomniacs. Furthermore, even if alerting drugs significantly improve MWT scores there is no data available concerning the impact of these drugs on fitness to drive. This lack of knowledge is a major handicap to evaluate driving skills of treated patients suffering from excessive daytime sleepiness. The main objective of our project is to test the predictive value of the MWT on real and simulated driving performances in untreated and treated sleepy patients suffering from narcolepsy and hypersomnia. Inclusion of healthy volunteers will allow to collect reference data about somnolence during MWT.

ELIGIBILITY:
Inclusion Criteria for Patients:

* Narcoleptic patients with or without cataplexy or hypersomniacs
* aged from 18 to 65 years,
* treated for attacks of cataplexy,
* treated with a maximum dose of Modiodal: 400 mg per day (4 tablets of 100mg),
* without any other disease which could be responsible of excessive daytime sleepiness,
* having their driver's licence,
* driving more than 5000 Km/year,
* registered to French national health and pensions organization,
* having regular timetables of life 7 days before beginning the study,
* having given their written light agreement in order to participate in the study.

Inclusion Criteria for Healthy Volunteers:

* without any sleep disorders,
* having their driver's licence since at least 2 years,
* driving more than 5000 Km/year,
* registered to French national health and pensions organization,
* having regular timetables of life 7 days before beginning the study,
* having given their written light agreement in order to participate in the study.

Exclusion Criteria for Patients:

* Night workers,
* breast-feeding or pregnant women
* Beck's scale score < 8,
* neurologic disease,
* cardiovascular disorders including cardiac arrhythmia,
* sleep disorders except narcolepsy and hypersomnia,
* pulmonary disorders,
* renal disorders,
* endocrinal disorders,
* having participated in a clinical study during the last 6 months,
* unable to drive.

Exclusion Criteria for Healthy Volunteers:

* Night workers,
* neurologic disease,
* cardiovascular disorders,
* sleep disorders,
* pulmonary disorders,
* renal disorders,
* endocrinal disorders,
* having participated in a clinical study during the last 6 months,
* unable to drive.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2010-03; Primary Completion 2012-07 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Sleep latency during MWT, number of vehicle's line crossing on the road, standard deviation of the vehicle's position on the road | for each condition, at day 4 for patients or day 1 for healthy volonteers

SECONDARY OUTCOMES:
Subjective sleepiness (Karolinska and VAS scales) | for each condition, at day 4 and 5 for patients or day 1 for healthy volonteers
nocturnal sleep quality and quantity will be measured by PSG and Actimetry. | For each condition, at day 4 and 5 for patients or day 1 for healthy volonteers

CONTACTS AND LOCATIONS:
Overall Officials: Pierre PHILIP, MD, PHD, Principal Investigator — University Hospital, Bordeaux
Locations (2):
- France (2):
  - GENNPHASS - CHU de Bordeaux, Bordeaux
  - AP-HP - Hôpital de l'Hôtel-Dieu, Paris

REFERENCES:
- [Background] Reyner LA, Horne JA, Reyner A. Gender- and age-related differences in sleep determined by home-recorded sleep logs and actimetry from 400 adults. Sleep. 1995 Feb;18(2):127-34. PMID 7792492
- [Background] Guilleminault C, Pelayo R, Leger D, Philip P, Ohayon M. Sleep-disordered breathing and upper-airway anomalies in first-degree relatives of ALTE children. Pediatr Res. 2001 Jul;50(1):14-22. doi: 10.1203/00006450-200107000-00006. PMID 11420413
- [Background] Philip P, Mitler M. Sleepiness at the wheel: symptom or behavior? Sleep. 2000 Jun 15;23 Suppl 4:S119-21. No abstract available. PMID 10893083
- [Background] Findley LJ, Unverzagt ME, Suratt PM. Automobile accidents involving patients with obstructive sleep apnea. Am Rev Respir Dis. 1988 Aug;138(2):337-40. doi: 10.1164/ajrccm/138.2.337. PMID 3195832
- [Background] Sleep apnea, sleepiness, and driving risk. American Thoracic Society. Am J Respir Crit Care Med. 1994 Nov;150(5 Pt 1):1463-73. doi: 10.1164/ajrccm.150.5.7952578. No abstract available.
- [Background] Barbe, Pericas J, Munoz A, Findley L, Anto JM, Agusti AG. Automobile accidents in patients with sleep apnea syndrome. An epidemiological and mechanistic study. Am J Respir Crit Care Med. 1998 Jul;158(1):18-22. doi: 10.1164/ajrccm.158.1.9709135. PMID 9655701
- [Background] Teran-Santos J, Jimenez-Gomez A, Cordero-Guevara J. The association between sleep apnea and the risk of traffic accidents. Cooperative Group Burgos-Santander. N Engl J Med. 1999 Mar 18;340(11):847-51. doi: 10.1056/NEJM199903183401104. PMID 10080847
- [Background] Lloberes P, Levy G, Descals C, Sampol G, Roca A, Sagales T, de la Calzada MD. Self-reported sleepiness while driving as a risk factor for traffic accidents in patients with obstructive sleep apnoea syndrome and in non-apnoeic snorers. Respir Med. 2000 Oct;94(10):971-6. doi: 10.1053/rmed.2000.0869. PMID 11059950
- [Background] Masa JF, Rubio M, Findley LJ. Habitually sleepy drivers have a high frequency of automobile crashes associated with respiratory disorders during sleep. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1407-12. doi: 10.1164/ajrccm.162.4.9907019. PMID 11029353
- [Background] Sagaspe P, Taillard J, Chaumet G, Guilleminault C, Coste O, Moore N, Bioulac B, Philip P. Maintenance of wakefulness test as a predictor of driving performance in patients with untreated obstructive sleep apnea. Sleep. 2007 Mar;30(3):327-30. PMID 17425229
- [Background] George CF, Boudreau AC, Smiley A. Effects of nasal CPAP on simulated driving performance in patients with obstructive sleep apnoea. Thorax. 1997 Jul;52(7):648-53. doi: 10.1136/thx.52.7.648. PMID 9246139
- [Background] Poceta JS, Timms RM, Jeong DU, Ho SL, Erman MK, Mitler MM. Maintenance of wakefulness test in obstructive sleep apnea syndrome. Chest. 1992 Apr;101(4):893-7. doi: 10.1378/chest.101.4.893. PMID 1555458
- [Background] Mitler MM, Walsleben J, Sangal RB, Hirshkowitz M. Sleep latency on the maintenance of wakefulness test (MWT) for 530 patients with narcolepsy while free of psychoactive drugs. Electroencephalogr Clin Neurophysiol. 1998 Jul;107(1):33-8. doi: 10.1016/s0013-4694(98)00044-3. PMID 9743270
- [Background] Meurice JC, Marc I, Series F. Efficacy of auto-CPAP in the treatment of obstructive sleep apnea/hypopnea syndrome. Am J Respir Crit Care Med. 1996 Feb;153(2):794-8. doi: 10.1164/ajrccm.153.2.8564134.
- [Background] Tiihonen M, Partinen M. Polysomnography and maintenance of wakefulness test as predictors of CPAP effectiveness in obstructive sleep apnea. Electroencephalogr Clin Neurophysiol. 1998 Dec;107(6):383-6. doi: 10.1016/s0013-4694(98)00079-0. PMID 9922082
- [Background] Randomized trial of modafinil for the treatment of pathological somnolence in narcolepsy. US Modafinil in Narcolepsy Multicenter Study Group. Ann Neurol. 1998 Jan;43(1):88-97. doi: 10.1002/ana.410430115. PMID 9450772
- [Background] Findley LJ, Suratt PM, Dinges DF. Time-on-task decrements in "steer clear" performance of patients with sleep apnea and narcolepsy. Sleep. 1999 Sep 15;22(6):804-9. doi: 10.1093/sleep/22.6.804. PMID 10505827
- [Background] Findley L, Unverzagt M, Guchu R, Fabrizio M, Buckner J, Suratt P. Vigilance and automobile accidents in patients with sleep apnea or narcolepsy. Chest. 1995 Sep;108(3):619-24. doi: 10.1378/chest.108.3.619. PMID 7656606
- [Background] Grubb TC. Narcolepsy and highway accidents. JAMA. 1969 Sep 15;209(11):1720. No abstract available. PMID 5820175
- [Background] Bartels EC, Kusakcioglu O. Narcolepsy: a possible cause of automobile accidents. Lahey Clin Found Bull. 1965;14(1):21-6. No abstract available. PMID 5828637
- [Background] Aldrich MS. Automobile accidents in patients with sleep disorders. Sleep. 1989 Dec;12(6):487-94. doi: 10.1093/sleep/12.6.487. PMID 2595172
- [Background] O'Hanlon JF, Volkerts ER. Hypnotics and actual driving performance. Acta Psychiatr Scand Suppl. 1986;332:95-104. doi: 10.1111/j.1600-0447.1986.tb08985.x. PMID 3554901
- [Background] Ramaekers JG, O'Hanlon JF. Acrivastine, terfenadine and diphenhydramine effects on driving performance as a function of dose and time after dosing. Eur J Clin Pharmacol. 1994;47(3):261-6. doi: 10.1007/BF02570506. PMID 7867679
- [Background] Philip P, Sagaspe P, Moore N, Taillard J, Charles A, Guilleminault C, Bioulac B. Fatigue, sleep restriction and driving performance. Accid Anal Prev. 2005 May;37(3):473-8. doi: 10.1016/j.aap.2004.07.007. PMID 15784201
- [Background] Philip P, Sagaspe P, Taillard J, Valtat C, Moore N, Akerstedt T, Charles A, Bioulac B. Fatigue, sleepiness, and performance in simulated versus real driving conditions. Sleep. 2005 Dec;28(12):1511-6. doi: 10.1093/sleep/28.12.1511. PMID 16408409
- [Background] Philip P, Taillard J, Moore N, Delord S, Valtat C, Sagaspe P, Bioulac B. The effects of coffee and napping on nighttime highway driving: a randomized trial. Ann Intern Med. 2006 Jun 6;144(11):785-91. doi: 10.7326/0003-4819-144-11-200606060-00004. PMID 16754920
- [Background] Mitler MM, Gujavarty KS, Browman CP. Maintenance of wakefulness test: a polysomnographic technique for evaluation treatment efficacy in patients with excessive somnolence. Electroencephalogr Clin Neurophysiol. 1982 Jun;53(6):658-61. doi: 10.1016/0013-4694(82)90142-0. PMID 6177511
- [Background] Sangal RB, Thomas L, Mitler MM. Maintenance of wakefulness test and multiple sleep latency test. Measurement of different abilities in patients with sleep disorders. Chest. 1992 Apr;101(4):898-902. doi: 10.1378/chest.101.4.898. PMID 1555459
- [Background] Lee KA, Hicks G, Nino-Murcia G. Validity and reliability of a scale to assess fatigue. Psychiatry Res. 1991 Mar;36(3):291-8. doi: 10.1016/0165-1781(91)90027-m. PMID 2062970
- [Background] Vallieres A, Morin CM. Actigraphy in the assessment of insomnia. Sleep. 2003 Nov 1;26(7):902-6. doi: 10.1093/sleep/26.7.902. PMID 14655927
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343